CLINICAL TRIAL: NCT03576287
Title: Apremilast as Anti-pruritic Treatment in Patients With Prurigo Nodularis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanja Todberg, MD (Other)
Responsible Party: Sponsor-Investigator, Tanja Todberg, MD, MD, principal investigator, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-003018-29
Record Dates: First submitted 2017-06-16; First posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Prurigo Nodularis
Keywords: apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apremilast (Experimental): apremilast standard doses
  Interventions: Drug: Apremilast Oral Product

INTERVENTIONS:
Drug: Apremilast Oral Product — Apremilast

SUMMARY:
This study will evaluate the anti-pruritic effect of apremilast in patients with known PN.

DETAILED DESCRIPTION:
Prurigo nodularis(PN) is a chronic skin disease, characterized by severe pruritus, multiple hyperkeratotic nodules and papules often located on the extensor part of the upper and lower extremities with a symmetrical distribution. The disease often appears between 20-60 years of age affecting men and women equally.

The pathogenesis of PN is poorly understood and it is unknown whether PN is a primary dermatological disease or if it arises secondary to intense pruritus and scratching of the skin with other diseases being the cause of the itching.

A number of studies have investigated if certain biochemical parameters are involved in mediating PN e.g. studies have indicated that the small nerve fibres in dermis in lesioned skin have an increased density of Substance P (neuropeptide and a well-known mediator of pruritus. when compared to non-lesioned skin.Other studies have suggested that patients with PN have a high presence of nerve growth factor (NGF) in dermis leading to modulation of the small nerve fibres, as well as an increased number of eosinophilic granulocytes, mast- and Merkel cells. Additionally, studies have found increased levels of IL-6 and IL-31 in blood in patient with PN. However the pathogenesis of PN remains unknown.

Among patients with atopic dermatitis there is a higher frequency of patients with PN as well as PN seem to be associated with certain liver- and kidney diseases. Anxiety and depression are also more common in patients with PN.

Patients with PN suffer from impaired quality of life due to ongoing pruritus and skin lesions(5). PN is mainly treated with topical steroids, UVB, PUVA or thalidomide, although none of these treatments seem to be able to control the disease and furthermore a number of these treatments are associated with several side effects.

As the phosphodiesterase 4 (PDE4)-inhibitor (apremilast) have shown a , it is speculated that apremilast may have an effect in patients with PN. Lack of effective treatments for PN supports further development for treatment options.

This study will evaluate the anti-pruritic effect of apremilast in patients with known PN. This interventional study, will be performed at the Department of Dermatology and Allergy at Herlev and Gentofte Hospital (Gentofte site), University of Copenhagen, Hellerup, Denmark.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* PN verified diagnosis by characteristic clinical features
* Moderate to severe PN
* Failure of local steroid and light treatment to control disease and symptoms.
* Be able to speak and understand Danish.
* Patients must have given their informed consent to the protocol and to the clinical procedures.

Exclusion Criteria:

* Patients who have received any local anti-inflammatory treatment 2 weeks prior to day 0
* Patients who have received any systemic anti-inflammatory treatment 4 weeks prior to day 0 or 5 pharmacokinetic half-lives, whichever is longer
* Patients who have received any other study medication 4 weeks prior to day 0
* Patients with other clinically significant disorders
* Patients with active TB/serious infections
* Any psychiatric condition which in the Investigators opinion would preclude the patient from adhering to the protocol or completing the study per protocol. Patients with previous endogene depression.
* Pregnancy
* Nursing
* Women of child-bearing potential must use effective contraception which includes IUD, oral, injected or implanted hormonal device, hormone patch, vaginal hormonal ring og sterilization.

  * Occlusive cap or condom with spermicidal cream is not considered as an effective contraception. Post-menopausal women (> 12 months of amenorrhea) are allowed not to use contraception.
* Patients who have received any live vaccines 6 weeks prior to day 0 or who are planning to receive a live vaccine during the study
* Allergy to apremilast or any of the other ingredients in Otezla®

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
1. Reduction in mean absolute VAS-pruritus score after 12 weeks treatment with apremilast compared to mean VAS-pruritus score before treatment with apremilast | 12 weeks
  1. Reduction in mean absolute VAS-pruritus score after 12 weeks treatment with apremilast compared to mean VAS-pruritus score before treatment with apremilast

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermato-Allergology, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No